CLINICAL TRIAL: NCT03578757
Title: Stress Management in Obesity During a Thermal Spa Residential Program: a Randomized Controlled Trial
Brief Title: Stress Management in Obesity During a Thermal Spa Residential Program
Acronym: ObesiStress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Regional Council of Auvergne-Rhône-Alpes (Other); European Regional Development Fund (Other); Spa resort of Vichy, Compagnie de Vichy, 1 et 3 avenue Eisenhower, 03200 Vichy, France (Unknown); Hospital of Vichy, Boulevard Denière, 03200 Vichy, France (Unknown); Université d'Auvergne (Other); LaPEC laboratory (EA 4278), Avignon University, Avignon, France (Unknown); Innovatherm (Industry); Center of Auvergne for Obesity and its health-related risks (CALORIS), Auvergne, France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHU-385; 2016 A01774 47 (Other: 2016 A01774 47)
Record Dates: First submitted 2018-03-26; First posted 2018-07-06 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Obesity; Stress
Keywords: stress; prevention; obesity; spa; psychology; biomarkers
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Masking Description: No masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): stress management program and the same usual practice (restrictive diet, physical activity and thermal spa treatment)
  Interventions: Behavioral: 21-day residential program
- usual practice group (Active Comparator): Both groups will benefit of a 21-day residential program at the thermal spa resort combining corrections of eating disorders
  Interventions: Behavioral: 21-day residential program

INTERVENTIONS:
Behavioral: 21-day residential program — Both groups will benefit of a 21-day residential program at the thermal spa resort combining corrections of eating disorders (and a negative energy balance of 500 kcal/day), physical activity (2h30 per day, minimum), thermal spa treatment (2h per day, minimum), and health education (1h30 per day, minimum: cooking, nutrition and physical activity classes…). Physical activity will be diverse (endurance, strength, circuit training) and personalized to the target of each participant.
  The intervention group will benefit from psychological interventions based on validated approaches of stress (3 x 1h30 per week). Participants will attend psychological sessions by group of less than 10 individuals. Individual meeting with the psychologist will occur at least twice: at the beginning of the residential program and at the end.
  After the spa residential program, participants will undergo a one-year at-home follow-up.

SUMMARY:
Stress can lead to obesity via inappropriate eating. In addition, obesity is a major stress factor. Furthermore, stressed people are also those who have the greatest difficulties to lose weight. The relationships between obesity and stress are biological via the action of stress on the major hormones regulating appetite (leptin, ghrelin). International recommendation proposals suggest to implement stress management programs in obesity for a sustainable weight loss. Moreover, stress and obesity are two public health issues. Among the multiple physical and psychological consequences of stress and obesity, increased mortality and cardiovascular morbidity seem the main concern. Many spa resorts are specialized in the treatment of obesity in France but actually no thermal spa proposes a specific program to manage stress in obesity.

The main hypothesis is that a thermal spa residential program (21 days) of stress management in obesity will exhibit its efficacy through objective measures of well-being and cardiovascular morbidity.

DETAILED DESCRIPTION:
The Obesi-Stress protocol was designed to provide a better understanding of the effect of a spa residential program combined with a stress management program on the improvement of heart rate variability in the treatment of obesity.

In the present protocol, parameters are measured on five occasions (inclusion, at the start of the spa, at the end of the spa, at 6 months and at 12 months).

Statistical analysis will be performed using Stata software (version 13; Stata-Corp, College Station, Tex., USA). All statistical tests will be two-sided and p<0.05 will be considered significant. After testing for normal distribution (Shapiro-Wilk test), data will be treated either by parametric or non-parametric analyses according to statistical assumptions. Inter-groups comparisons will systematically be performed 1) without adjustment and 2) adjusting on factors liable to be biased between groups.

Analysis will be performed using Student t-test or Mann-Whitney tests. Linear regression (with logarithmic transformation if necessary) considering an adjustment on covariates fixed according to univariate results, epidemiological relevance and observance to physical activity will complete the analysis. Comparisons of categorical variables will be performed using Chi-squared or Fischer test. Relations between quantitative outcomes will be analyzed using correlation coefficients (Pearson or Spearman). Fisher's Z transformation and William's T2 statistic will be performed to compare correlations between variables and within a single group of subjects. Longitudinal data will be treated using mixt-model analyses in order to treat fixed effects group, time and group x time interaction taking into account between and within participant variability.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese participants with Body Mass Index (BMI) >25 kg.m-2
* Spontaneously candidate to the spa program of Vichy for management of obesity
* Aged over 18 years old
* A stable weight during the last three months
* No hepatic, renal or endocrine diseases uncontrolled
* Ability to give a written informed consent -- Affiliated to French health care system (for France)

Exclusion Criteria:

* Participant refusal to participate
* Pregnant and breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
heart rate variability (biomarker of both stress and morbidity/mortality) | HRV changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year.
  To assess the ability of a short spa residential program of management of work-related stress in increasing heart rate variability, a biomarker of both stress and morbidity/mortality.
  Heart rate variability will be measured by zephyr during 26h recording time

SECONDARY OUTCOMES:
skin conductance | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year.
  skin conductance will be measured using Wirst band electrodes
blood flow velocity | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year
  blood flow velocity will be measured using laser speckle contrast imaging
myocardial longitudinal strain | Changes overtime is being assessed. Outcomes will be measured at the beginning of the spa program (day 0) and at six months
  myocardial longitudinal strain will be measured using speckle tracking echocardiography
Genetic polymorphisms related to stress | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year
  Genetic polymorphisms related to stress will be measured using blood cells (angiotensin converting enzyme and serotonin)
Demographics information | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year.
  Demographics information will be obtained using a single questionnaire including questions on age, gender, qualification, personal work status, ethnicity, life and occupational events
Anthropometry | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year
  Anthropometry parameters will be obtained according to the ISAK recommendations
Body composition | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year
  Body composition (muscle and fat) will be measured using Impedancemeter
Body composition | Changes overtime is being assessed. Outcomes will be measured at the beginning of the spa program (day 0) and at one year
  Body composition (muscle and fat) will be measured using dual x-ray absorption
bone microarchitecture | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year.
  bone microarchitecture will be measured using peripheral quantitative computed tomography
bone mass | Changes overtime is being assessed. Outcomes will be measured at the beginning of the spa program (day 0) and at one year.
  bone mass will be measured using dual x-ray absorption
bone mass | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year.
  bone mass will be measured using quantitative ultrasounds
General Health | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year.
  General Health will be measured using the General Health Questionnaire, (there is no score, just informative health information)
Physical Activity | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year.
  Physical Activity will be measured using the Recent Physical Activity Questionnaire (All activities are categorised depending on intensity: sedentary (<1.5 MET); light (1.5 to <3 MET), moderate-to-vigorous (>3MET))Questionnaire
Depression and anxiety | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year
  Depression and anxiety will be measured using the Hospital anxiety and depression scale (scale range from 0 to 3, with a total score between 0 to 21. Threshold score is 8
Burn-out | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year.
  Burn-out will be measured using the Maslach Burn Out Inventory (scale range from 0 to 6, with 0 = never and 6 = almost always)
Job content | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year
  Job content will be measured using the Karasek questionnaire (scale range from 1 to 4, with 1= not agreed and 4 = totally agreed)
anxiety | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year
  anxiety will be measured using the state and trait anxiety inventory scale (scale range from 1 to 4, with a total score between 20 to 80. If <35 poor level of anxiety, if > 66 very high level of anxiety)
mindfulness | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year.
  mindfulness will be measured using the Freiburg mindfulness inventory scale (scale range from 1 to 4, with 1 = almost never, 4 = almost always)
self-efficacy | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year
  self-efficacy will be measured using the perceived self-efficacy scale (scale range from 1 to 4, with 1= wrong and 4 = true)
Alexithymia | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year
  Alexithymia will be measured using the Toronto Alexithymia scale (scale range from 1 to 5, with 1 = not agreed, 5 = totally agreed)
coping responses | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year
  coping responses will be measured using the brief COPE questionnaire (scale range from 1 to 4, with 1 = not agreed, 4 = totally agreed)
emotion regulation | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year.
  emotion regulation will be measured using the emotion regulation questionnaire (scale range from 1 to 7, with 1 = not agreed, 7 = totally agreed)
metacognition | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year
  metacognition will be measured using the metacognition questionnaire MQC-30 (scale range from 1 to 4, with 1 = not agreed, 4 = totally agreed)
illness perception | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year
  illness perception will be measured using the brief illness perception questionnaire (B-IPQ 9 items, scale range from 0 to 10)
lifestyle behaviours | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year
  lifestyle behaviours will be measured using the lifestyle questionnaire
workplace stress | : Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year.
  workplace stress will be measured using the Inner Correspondence/Peaceful Harmony with practices - ICPH (17 items, a 5-point scale from disagreement to agreement, scores >50% indicate higher agreement while scores <50 indicate disagreement).
Basic biology | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year.
  HbA1c (mmol/mol) will be measured using endocrine assays
appetite markers | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year.
  Leptin (ng/mL) will be measured using endocrine assays
Pro-inflammatory cytokine | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year
  IL-1β will be measured using endocrine assays
Telomeres length | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year
  Telomeres length will be measured using endocrine assays
stress markers | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year.
  Cortisol (nmol/l) will be measured using endocrine assays
adrenal function | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year.
  adrenal function will be measured using endocrine assays (Dehydroepiandrosterone - DHEAS)
neurotrophic factors | Changes overtime is being assessed. Outcomes will be measured at inclusion, at the beginning of the spa program (day 0), day 21, at six months and at one year.
  neurotrophic factors will be measured using endocrine assays (Brain-Derived Neurotrophic Factor -BDNF)

CONTACTS AND LOCATIONS:
Overall Officials: Frederic DUTHEIL, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Dutheil F, Chaplais E, Vilmant A, Courteix D, Duche P, Abergel A, Pfabigan DM, Han S, Mobdillon L, Vallet GT, Mermillod M, Boudet G, Obert P, Izem O, Miolanne-Debouit M, Farigon N, Pereira B, Boirie Y. Stress management in obesity during a thermal spa residential programme (ObesiStress): protocol for a randomised controlled trial study. BMJ Open. 2019 Dec 23;9(12):e027058. doi: 10.1136/bmjopen-2018-027058. PMID 31874865